CLINICAL TRIAL: NCT04333823
Title: Adolescent Type 1 Diabetes Treatment With SGLT2i for hyperglycEMia & hyPerfilTration Trial
Acronym: ATTEMPT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Farid Mahmud, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO1940
Record Dates: First submitted 2020-03-30; First posted 2020-04-03 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Dapagliflozin; Type 1 Diabetes; Adolescent; Hyperfiltration; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: 1:1 ratio for treatment with Dapagliflozin or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Dapagliflozin) (Experimental): Dapagliflozin 5mg tablet taken by mouth once daily for 16 weeks
  Interventions: Drug: Dapagliflozin 5mg
- Control (Placebo) (Placebo Comparator): Dapagliflozin 5mg tablet taken by mouth once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 5mg — Dapagliflozin tablet
  Other Names: FORXIGA 5mg; ATC Code: A10BK01; DIN: 02435462
  Arms: Intervention (Dapagliflozin)
Drug: Placebo — Sugar pill manufactured to mimic Dapagliflozin 5mg tablet
  Other Names: Placebo (for Dapagliflozin)
  Arms: Control (Placebo)

SUMMARY:
The ATTEMPT (Adolescent Type 1 diabetes Treatment with SGLT2i for hyperglycEMia & hyPerfilTration Trial) is a multi-center, double-blinded, randomized, placebo-controlled trial to evaluate the effect of treatment with Dapagliflozin when compared to placebo, in combination with adjustable insulin, on measured GFR in adolescents with T1D 12 to <19 years of age over a 16-week treatment period.

DETAILED DESCRIPTION:
The ATTEMPT (Adolescent Type 1 diabetes Treatment with SGLT2i for hyperglycEMia & hyPerfilTration Trial) is designed to evaluate the impact of Dapagliflozin versus placebo in combination with insulin therapy. This trial will assess detailed renal mechanistic evaluations, with direct measurement of GFR, to understand the important physiologic impacts of SGLT2 inhibition on the early onset manifestations and progression of diabetes complications within this age group.

Fundamentally, the ATTEMPT trial will provide essential information in establishing a framework for this young cohort to evaluate key physiologic, mechanistic and metabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to consent; participants or their parents/legal guardians or responsible representatives must be willing and able to give signed informed consent. Participants without capacity must provide assent where applicable.
2. Diagnosis of Type 1 Diabetes, defined by American Diabetes Association Criteria, for at least 12 months.
3. Sex: Male and Female.
4. Age: 12 years to <19 years.
5. HbA1c: 7.0-10 % at time of screening. Participants with a lower (6.5 to <7.0%) or a higher HbA1c (>10.0 to 11.0%) may be considered, based upon investigator discretion, if patient is adherent with study safety criteria, including a good understanding of diabetes management, regular and consistent blood glucose monitoring, appropriate ketone testing and DKA symptom recognition, appropriate adjustment of insulin doses for meals and activity as well as illness.
6. On Insulin Therapy: Daily injections, to include TID (three times a day), multiple daily dose insulin injection (MDI, > 3 injections daily) or Pump (CSII).
7. A minimum total daily dose (TDD) of insulin ≥0.6 Units/kilogram/day.
8. Females of child bearing potential must be willing to use medically acceptable contraception for the duration of the study and at least one week plus 30 days (one menstrual cycle) post last dose of study drug.

Exclusion Criteria:

1. Pregnancy (positive serum or urine pregnancy test) or breastfeeding.
2. Allergies to any member of SGLT2i class of medications.
3. Type 2 diabetes, Maturity onset Diabetes of Young (MODY) as defined by American Diabetes Association Criteria or pancreatic disorders with resultant impaired pancreatic function.
4. Body Mass Index > 99.9th percentile by age and sex.
5. Presence of severe hypoglycemic event requiring assistance or glucagon rescue medication within 30 days of screening visit.
6. Presence of documented Diabetic Ketoacidosis (DKA) within 90 days of screening visit.
7. Current and/or anticipated adoption of a carbohydrate-restrictive diet
8. Current eating disorder or weight loss >10% of body weight within 90 days of screening visit.
9. Current and or/anticipated systemic corticosteroid therapy for greater than 5 days (not including inhaled, topical, eye or ear drops containing corticosteroids).
10. Current or history of alcohol, drug or substance abuse.
11. Participation in another drug intervention study within the past 30 days.
12. Presence of a clinically untreated or unstable medical condition (including diagnosed Hypertension, SBP>95%) or laboratory finding that may interfere with any aspect of the study.
13. Any concomitant medication known to interfere with the investigational product and/or renal function and/or planned study assessments based on investigators' judgement.
14. Unable to adhere with study safety criteria, in the investigator's opinion, including a suboptimal understanding of diabetes management that would include regular and consistent blood glucose monitoring, appropriate ketone testing and DKA symptom recognition, appropriate adjustment of insulin doses for meals and activity as well as illness
15. Participants are not allowed to change their insulin administration method (injection to pump or vice versa) throughout the study period, nor change to hybrid or closed loop insulin pumps during the study period.
16. Known Hypersensitivity to Iohexol

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Measured Glomerular Filtration Rate (mGFR) | 16 weeks
  Change in mGFR from baseline to the end of the 16-week treatment period.

SECONDARY OUTCOMES:
Glycated Hemoglobin A1c (HbA1c) | 16 weeks
  Change in HbA1c from baseline to the end of the 16-week treatment period.
Adverse events | 16 weeks
  Rate of adverse events reported from baseline to the end of the 16-week treatment period.
Diabetes Ketoacidosis (DKA) | 16 weeks
  Rate of confirmed DKA events from baseline to the end of the 16-week treatment period. All reported and suspected DKA events will be reviewed for confirmation by the study's DKA Adjudication Committee.
Hypoglycemic events | 16 weeks
  Rate of hypoglycemic events requiring assistance from baseline to the end of the 16-week treatment period.
Urinary and Genitourinary Tract Infections | 16 weeks
  Rate of urinary and genitourinary tract infections reported from baseline to the end of the 16-week treatment period.
Blood Glucose Profile | 16 weeks
  Change in ambulatory glucose profiles (AGP) from pre-drug initiation to the end of the 16-week treatment period.
Glycemic Variability | 16 weeks
  Change in time-in-range (TIR) from baseline to the end of the 16-week treatment period as measured by CGM. TIR is defined as the proportion of time (in %) spent with blood glucose levels between 3.9 and 10.0 mmol/L and will be determined using CGM.
Weight | 16 weeks
  Change in body weight (in kg) from baseline to the end of the 16-week treatment period.
Body Mass Index (BMI) | 16 weeks
  Change in Body Mass Index in (kg/m<sup>2</sup>) from baseline to the end of the 16-week treatment period.
Maturation | 16 weeks
  Assessed by Tanner pubertal staging at baseline and the end of the 16-week treatment period.
Total Daily Insulin Dose (TDID) | 16 weeks
  Change in the total daily dose of insulin (in IU) from baseline to the end of the 16-week treatment period.

OTHER OUTCOMES:
Flow-Mediated Dilation (FMD) | 16 weeks
  Change in flow mediated dilation using high resolution ultrasound from baseline to the end of the 16-week treatment period.
Pulse Wave Velocity (PWV) | 16 weeks
  Change in pulse pressure waveforms from baseline to the end of the 16-week treatment period.
Heart Rate Variability (HRV) | 16 weeks
  Change in heart rate variability from baseline to the end of the 16-week treatment period.
Caloric Intake | 16 weeks
  Change in daily caloric intake (in kcals) from baseline to the end of the 16-week treatment period.
Macronutrient Intake | 16 weeks
  Change in daily macronutrient intake (carbohydrates, fat, protein) in grams per kcals from baseline to the end of the 16-week treatment period.
Treatment Satisfaction | 16 weeks
  Assessed using the Diabetes Treatment Satisfaction Questionnaire (DTSQ), using a standardized scoring system.
Diabetes Management | 16 weeks
  Assessed using the Diabetes Management Questionnaire (DMQ) using a 20 item questionnaire with standardized scoring.
BOLD MRI | 16 weeks
  Changes in functional renal imaging
Exercise Session - Blood Glucose Levels | 4 weeks
  Change in blood glucose levels from pre- to post-exercise from baseline to 4 weeks post-drug initiation. Participants in the optional exercise component will undergo a moderate activity exercise session and will have their blood tested before and at the end of the 60-minute session.
Exercise Session - Blood Glucose Variability | 4 weeks
  Change in time-in-range (TIR) during a moderate activity exercise session from baseline to 4 weeks post-drug initiation. TIR is defined as the proportion of time (in %) spent with blood glucose levels between 3.9 and 10.0 mmol/L and will be determined using CGM.

CONTACTS AND LOCATIONS:
Overall Officials: Farid H Mahmud, MD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Children's Hospital Colorado Anschutz Medical Campus, Aurora, Colorado, United States
- Canada (2):
  - London Health Sciences Centre Children's Hospital, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmud FH, Bjornstad P, Clarson C, Clarke A, Anthony SJ, Curtis J, Elia YT, McArthur L, Mertens L, Moineddin R, Kirsch S, Coles N, Maione M, Furman M, Babalola F, Tommerdahl KL, Harrington J, Riddell MC, Prasad P, Huang L, Heerspink HJL, Cherney DZI. Adjunct-to-insulin therapy using SGLT2 inhibitors in youth with type 1 diabetes: a randomized controlled trial. Nat Med. 2025 Jul;31(7):2317-2324. doi: 10.1038/s41591-025-03723-6. Epub 2025 Jun 6. PMID 40481206